CLINICAL TRIAL: NCT06884605
Title: The Effect of Problem-Based Learning and Mind Mapping Method on Identifying Nursing Interventions
Brief Title: Problem-Based Learning and Mind Mapping Method
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 12
Record Dates: First submitted 2025-03-11; First posted 2025-03-19 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-03

CONDITIONS: Nursing Education
Keywords: problem-based learning; mind mapping; nursing intervention; nursing students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nursing students: problem-based learning and mind mapping

SUMMARY:
Problem-based learning and mind mapping methods contribute positively to the learning of nursing students and also improve their critical thinking skills.

DETAILED DESCRIPTION:
This study focuses on determining nursing interventions, which is an important stage of the nursing process. It is aimed to evaluate the effect of problem-based learning and mind mapping method on determining nursing interventions in nursing students. The research is original in its field in terms of using problem-based learning and mind mapping method simultaneously and focusing on nursing interventions. Therefore, the study is expected to be guiding for teaching staff as well as measuring the effect of nursing students on planning knowledge and nursing interventions.

ELIGIBILITY:
Inclusion Criteria:

* Not having received training on determining the nursing process and nursing interventions before
* Attending classes, attending post-test and follow-up tests

Exclusion Criteria:

* Having previously received training to determine the nursing process and nursing interventions
* Being absent from class, not attending the post-test and follow-up test

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Nursing students
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-05-05 (Actual)

PRIMARY OUTCOMES:
The effect of learning method on students' knowledge level | 03/10/2025-05/07/2025
  nursing students and educational methods
The effect of learning method on students' skill level | 03/10/2025-05/07/2025
  educational methods

CONTACTS AND LOCATIONS:
Overall Officials: Aysun Acun, PhD, Study Director — Bilecik Seyh Edebali Universitesi
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)